CLINICAL TRIAL: NCT06830746
Title: A Stylet-Driven ICD Lead Intended for Conduction System Pacing IDE Study
Brief Title: ASCEND CSP IDE Study
Acronym: ASCEND CSP IDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10549
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure; Ventricular Arrythmia
Keywords: ICD; CRT-D; LBBAP; conduction system pacing; lead
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Subjects undergoing ICD/CRT implant will be implanted with the CSP ICD Lead in the LBBAP location and undergo required electrical testing
  Interventions: Device: LBBAP Implant with a CSP ICD Lead

INTERVENTIONS:
Device: LBBAP Implant with a CSP ICD Lead — Required electrical testing for pacing, sensing, impedance and defibrillation will be completed

SUMMARY:
This is a prospective, multi-center, global, single-arm, pivotal investigational study designed to evaluate the safety and effectiveness of the CSP ICD Lead in a subject population indicated for ICD or CRT-D therapy.

The clinical investigation will enroll up to 414 subjects at up to 70 participating centers from the United States, Canada, Europe, and Asia Pacific.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must meet current clinical practice guidelines for implantation of ICD or CRT-D and will undergo one of the following:

   1. de novo Abbott ICD system implant (single or dual chamber)
   2. de novo Abbott CRT-D system implant and is intended to also undergo left ventricle coronary sinus lead implant (for patients indicated for CRT-D according to locally approved indications)
2. Subject is ≥ 18 years of age or age of legal consent, whichever age is greater.
3. Subject is willing to undergo implant defibrillation testing if requested. Subjects with AF in whom defibrillation testing is required must have been on or willing to be on uninterrupted anticoagulation therapy before, during, and after the implant procedure.
4. Subject is willing to comply with clinical investigation procedures and agrees to return to clinic for all required follow-up visits, tests, and exams.
5. Subject has been informed of the nature of the clinical investigation, agrees to its provisions and has provided a signed written informed consent, approved by the IRB/EC.

Exclusion Criteria:

1. Subject has had myocardial infarction or unstable angina within 40 days prior to signing consent
2. Subject has had recent cardiac revascularization (angioplasty, stent or bypass graft) in the 4 weeks prior to signing consent or planned within 3 months following consent
3. Subject has had any other therapeutic cardiovascular procedure (such as transcatheter aortic valve replacement, MitraClip, cardiac surgery, left atrial appendage closure, patent foramen ovale closure, or any ablation procedures) in the 3 months prior to signing consent or planned within 3 months following consent
4. Subject has had a recent Cerebrovascular Accident (CVA) or Transient Ischemic Attack (TIA) within 3 months of prior to signing consent
5. Subject has a life expectancy of less than 12 months
6. Subject has contraindications for standard RV transvenous and/or LBBAP lead placement (e.g., mechanical right heart valve)
7. Subject is contraindicated for ≤1mg Dexamethasone sodium phosphate.
8. Subject is pregnant or breastfeeding women, or women of childbearing potential and who are not on a reliable form of birth regulation method or abstinence
9. Subject has an existing pacemaker (including a temporary pacing system), ICD, CRT, or cardiac contractility modulation (CCM) device or leads
10. Subject has any evidence of active infection or undergoing treatment for an infection
11. Subject is enrolled or planning to enroll in another clinical trial that might confound the results of the present study
12. Subject has moderate or severe aortic stenosis
13. Subject has ventricular septal defect (VSD) or had prior surgery on the interventricular septum that could impact LBBAP implant, such as septal myomectomy, ethanol septal ablation, VSD repair, etc
14. Subject has end-stage renal disease
15. Subject has NYHA IV classification
16. Subject has undergone cardiac transplantation or have a classification of Status 1 for cardiac transplantation or consideration for transplantation during the study follow-up period
17. Subject has had previously extracted leads
18. Subject has had an LV Assist Device
19. Subject has had a failed LBBAP lead implant

Defibrillation testing exclusion criteria (these are part of general exclusion criteria when defibrillation testing is requested):

1. Subject has pre-existing or suspected pneumothorax during implant
2. Subject has current known intracardiac left atrial or Left Ventricular thrombus
3. Subject has severe proximal three-vessel or left main coronary artery disease without revascularization
4. Subject has Ejection Fraction less than 20%
5. Subject has recent stroke or transient ischemic attack (within the last 6 months)
6. Subject has known inadequate external defibrillation
7. Subject has any other known medical condition not listed that precludes their participation in the opinion of the investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 3 months post-implant
  Freedom from CSP ICD Lead-related Serious Adverse Device Effects (SADEs) through 3 months post-implant for subjects in which the CSP ICD Lead implant was attempted
Primary Effectiveness Endpoint 1 | 3-months post-implant
  3-month composite success rate of acceptable pacing capture thresholds and R-wave sense amplitudes of the CSP ICD Leads in the subjects with the CSP ICD Lead implanted at the LBBA
Primary Effectiveness Endpoint 2 | at implant
  Success rate of the defibrillation testing at implant in the subjects who complete the defibrillation test with the CSP ICD Lead implanted at the LBBA

CONTACTS AND LOCATIONS:
Locations (36):
- United States (15):
  - Heart Center Research LLC, Huntsville, Alabama
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Premier Cardiology, Inc., Newport Beach, California
  - University of California at San Diego (UCSD) Medical Center, San Diego, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - AdventHealth Orlando, Orlando, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Australia (4):
  - The Prince Charles Hospital, Chermside, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
- MUHC- Montreal General Hospital, Montreal, Canada
- France (3):
  - CHRU Hopital de Pontchaillou, Rennes, Brittan
  - CHU Trousseau, Chambray-lès-Tours, Centre-Val de Loire
  - Hôpital Pitié Salpetrière, Paris, Ile
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- India (3):
  - Max Super Specialty Hospital, New Delhi, National Capital Territory of Delhi
  - Sree Chitra Tirunal Institute for Medical Sciences & tech., Trivandrum, New Delhi
  - Velammal Medical College Hospital, Madurai, Tmlnadu
- Italy (2):
  - Ospedale S.S. Annunziata, Taranto, Apulia
  - Ospedale Niguarda Ca'Granda, Milan, Lombard
- Singapore (3):
  - National Heart Centre Singapore, Singapore, Singapore
  - Changi General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- Spain (2):
  - Hospital Universitari i Politècnic La Fe, Valencia, Valencia
  - Hospital Universitario Virgen de las Nieves, Granada
- Hopital Cantonal Universitaire de Geneva, Geneva, Canton of Geneva, Switzerland